CLINICAL TRIAL: NCT04909710
Title: Feasibility of Mobile Game System for Potential Treatment of Developmental Delays
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: we are suspending this study until we have continued funding.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Dennis Paul Wall, Associate Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB 39562
Record Dates: First submitted 2021-05-13; First posted 2021-06-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: digital; mobile; autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: The investigators will use parallel assignment to compare the device feasibility across children with autism and neurotypical children, who will serve as controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autism Case Group (Experimental): Autistic participants will receive mobile game system for 12 weeks and be asked to play a minimum of ten 90-second game sessions per week per child over 12 weeks. Research team will further require that at least three of these 10 weekly sessions with each child be with game decks displaying emotion.
  Interventions: Other: Mobile Game System for Potential Treatment of Developmental Delays
- Neurotypical Sibling Control Group (Other): Neurotypical control participants will receive the same mobile game system for 12 weeks and be asked to play a minimum of ten 90-second game sessions per week per child over 12 weeks. Research team will further require that at least three of these 10 weekly sessions with each child be with game decks displaying emotion.
  Interventions: Other: Mobile Game System for Potential Treatment of Developmental Delays

INTERVENTIONS:
Other: Mobile Game System for Potential Treatment of Developmental Delays — Mobile game system meant to generate valuable data for measuring progress and building novel artificial intelligence models while delivering impactful education for and treatment of children with developmental delays such as autism.

SUMMARY:
The investigators will test the feasibility and preliminary efficacy of a Mobile game system meant to generate valuable data for measuring progress and building novel artificial intelligence models while delivering impactful education for and treatment of children with developmental delays such as autism. Investigators will enroll children with autism aged 2-8 years old and their neurotypical sibling or an unrelated neurotypical control (aged 2-8 years old).

ELIGIBILITY:
Inclusion Criteria:

1. Parent or primary caregiver over 18 of a child with autism, we will enrich for children between the ages of 2 and 8 years old.
2. Autism diagnosis confirmed by a screener such as the Mobile Autism Risk Assessment (MARA) and or similar published tools.

Exclusion Criteria:

(1) Physical, intellectual, language related, or environmental limitations that prevent the ability for the family to play the game as intended.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in parent reported socialization subscale scores of the Vineland Adaptive Behavior Scales,2nd Edition (VABS-2) from baseline to week 12 Vineland Adaptive Behavior Scales, 2d edition (VABS-2) Socialization subscale of the Parent/Caregiver | Baseline (Week 0), Week 12
  The socialization subscale is up to 113 items, where raw scores are converted to Intelligence Quotient (IQ) type standard scores--v-scale scores (M=15, SD=3) where scores range from 1 to 24, and factor in age equivalents, growth scale values, and higher scores indicate better adaptive functioning.
Mobile Application Usage-Total games started. | Week 12
  App usage data by participants (children) comprised of total number of MojiMatch plus Charades Games started.

SECONDARY OUTCOMES:
Change in parent reported social responsiveness from week 0 to week 12 | Baseline (Week 0), Week 12
  The Social Responsiveness Scale-2 is a 65-item measure where parents rate their child selecting responses on a Likert Scale. This measure will be used to measure and identify social impairment associated with Autism Spectrum Disorder (ASD) and to quantify its severity Social Responsiveness Scale (SRS) raw scores measure social abilities with lower scores indicating better social skills. (Raw Score Range: 0 - 195 and T-Score Range: 37- above 90).
Change in mobile autism risk assessment score from week 0 to week 12 | Baseline (Week 0), Week 12
  A level 2 screening tool that has been validated in several studies and that uses a brief parent questionnaire with a 2 minute home video to generate a classification score that indicates severity of the autism phenotype (ranging from no autistic symptoms to severe autism) as well as confidence in the classification.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis P Wall, PhD, Principal Investigator — Associate Professor
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 1 year after study completion